CLINICAL TRIAL: NCT00545792
Title: A Pilot Study Evaluating The Safety Of Avastin And Pelvic Radiation In Women With Pelvic-Confined Recurrence of Gynecological Cancers
Brief Title: Safety Study Of Avastin And Pelvic Radiation In Women With Recurrent Gynecological Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Lowell General Hospital (Other); Saint Anne's Hospital (Other)
Responsible Party: Principal Investigator, Paul Nguyen, MD, Paul Nguyen MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-042; AVF3998s (Other: Genentech)
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Cervical Cancer; Endometrial Cancer; Ovarian Cancer; Vaginal Cancer; Carcinoma of the Vulva
Keywords: Recurrent Endometrial cancer; Recurrent Cervical cancer; Recurrent Ovarian cancer; Recurrent Vaginal cancer; Recurrent Vulvar cancer; Vaginal recurrence; Brachytherapy; Radiation Treatment; External Beam Radiation; Avastin; Bevacizumab
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin (Experimental): Avastin
  Interventions: Drug: Avastin

INTERVENTIONS:
Drug: Avastin — Avastin will be administered intravenously (vein) at 10mg/kg every two weeks starting day 1 for a total of 3 doses.
  Other Names: Bevacizumab

SUMMARY:
This research study is evaluating a drug called avastin in combination with standard radiation as a possible treatment for treatment for recurrent pelvic-confined gynecological cancer (i.e. endometrial, cervical, vulvar, ovarian or vaginal cancers).

DETAILED DESCRIPTION:
The purpose of this research study is to learn the effects (good and bad) of an antiangiogenic therapy drug (drugs that stop new blood vessel growth and starve a tumor by cutting off its blood supply) called avastin. Avastin is an antibody directed against vascular endothelial growth factor, or VEGF. VEGF is a potent, specific growth factor with a well-defined role in normal and abnormal blood vessel formation. It is present in a wide variety of normal tissues, but is produced in excess by most solid cancers (tumors). In the setting of cancer, VEGF promotes the growth of blood vessels that bring nutrients to tumor cells. In laboratory studies, avastin has been shown to inhibit the growth of several different types of human cancer cells.

This drug has been studied in at least 3500 people with breast, colorectal, renal, ovarian and lung cancer. It has not been studied in combination radiation therapy in people with recurrent gynecological cancer.

Previous clinical trials involving the use of avastin in combination with standard radiation in colorectal and pancreatic cancer show no significant increase in toxicity as compared to standard radiation therapy toxicity.

The primary objective of this study is to assess the toxicity of administering avastin with radiation for recurrent gynecological cancer. The secondary endpoint will be to assess the time to progression of the disease. This means we hope this treatment program will delay any regrowth of your cancer as compared to standard therapy with radiotherapy alone. In addition, how well you respond to the treatment, patterns of remission or recurrence will be measured.

ELIGIBILITY:
Inclusion Criteria:

* All patients (age > 18 years) will have locally recurrent gynecological cancer with a component of disease that will fit within a standard RT portal at the time of presentation
* ECOG performance status score 0-1
* All patients will have had a prior hysterectomy
* Histological confirmation of recurrent gynecological cancer, including adenocarcinoma, papillary serous carcinoma, clear cell carcinoma, or carcinosarcoma
* Age > 18 years
* Radiologic work-up computer tomography of the chest and abdomen, and computer tomography or MR of the pelvis confirming pelvis-confined recurrence
* Adequate renal function as evidenced by serum creatinine < 1.5 mg/dL
* Adequate hepatic function as evidenced by:

Serum total bilirubin < 1.5 mg/dL SGOT/SGPT < 3X the ULN for the reference lab

* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with a prior history of full course external beam radiation therapy to the pelvis (patients with prior vaginal brachytherapy may be included)
* Inability to comply with study and/or follow-up procedures
* Life expectancy of less than 12 weeks
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored avastin cancer study
* Known CNS disease (including history of encephalitis, multiple sclerosis or seizure disorder), except for treated brain metastasis
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Known CNS disease (including history of encephalitis, multiple sclerosis or seizure disorder)
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Any surgical procedure requiring an incision, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for any surgical procedure requiring an incision during the course of the study (excluding vascular access device placement or procedures that do not require an incision)
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either Urine protein:creatinine (UPC) ratio ≥ 1.0 at screening OR Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of avastin
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to give informed consent or cooperate and participate in the study or to interfere with the investigator's ability to interpret the results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-05; Primary Completion 2010-11 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Nguyen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Viswanathan AN, Lee H, Berkowitz R, Berlin S, Campos S, Feltmate C, Horowitz N, Muto M, Sadow CA, Matulonis U. A prospective feasibility study of radiation and concurrent bevacizumab for recurrent endometrial cancer. Gynecol Oncol. 2014 Jan;132(1):55-60. doi: 10.1016/j.ygyno.2013.10.031. Epub 2013 Nov 4. PMID 24201015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was between 2008-2010. Patients seen in consultation in a gynecologic oncology or radiation oncology clinic at any of the participating institutions and recommended to undergo radiation for recurrent gynecological cancer were evaluated for eligibility.
Pre-assignment Details: Pretreatment evaluations included medical interview, blood pressure check, complete blood count, chemistries, urine analysis and liver function tests. Tumor biopsy was performed at diagnosis. Radiologic imaging (CT, PET-CT, or MR) was performed at diagnosis.
Groups:
- Avastin: Avastin and daily radiation
  Avastin : Avastin will be administered intravenously (vein) at 10mg/kg every two weeks starting day 1 for a total of 3 doses.
Period: Overall Study
Arm/Group | Avastin
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Modified intention to treat (ITT), i.e., include all subjects that received and completed treatment.
Arm/Group | Avastin
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Toxicity Rates of Patients Treated With Concurrent Avastin and Daily Pelvic Radiation With no Other Concurrent Chemotherapy
Description: Toxicity was the cumulative number of events, all grades and categories, related to side effects from avastin and radiation including, but not limited to, bowel, bladder, skin, gynecologic and other morbidity.
Time Frame: 1-year
Population: 20 patients received and completed treatment.
Measure: Number; unit: Events
Arm/Group | Avastin
Number analyzed (Participants) | 20
Events | 766

2. Secondary Outcome: Single Point Estimate of 1-year Progression-free Survival of Patients Treated With Concurrent Avastin and Daily Pelvic Radiation With no Other Concurrent Chemotherapy
Description: Progression free survival was calculated from the date of diagnosis to the date of disease progression as detected by clinical examination or imaging.
Time Frame: 1-year
Population: 20 patients received and completed treatment.
Measure: Number; unit: participants
Arm/Group | Avastin
Number analyzed (Participants) | 20
participants | 16
Statistical Analysis 1: Comparison: Avastin; Single-arm feasibility study; Kaplan Meier analysis was applied to estimate one-year PFS distribution as well as to calculate proportion of patients remain progression free by month 12; Test type: Superiority or Other; Single point estiamte of 1-yr PFS = 0.8, 95% CI 2-sided [0.56 to 0.94] — The reported 1-year PFS rate 80% (Exact 95% CI: 56% - 94%) was the proportion of the patients remained progression free after 12 months

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Avastin
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin (N=20)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) — Grade 4
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
Portal Vein Flow (Vascular disorders) | 1 (1)
Hemorrhage, GI (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin (N=20)
Diarrhea (Gastrointestinal disorders) | 18 (42)
Vascular event (Vascular disorders) | 1 (2)
Genitourinary/bladder event (Renal and urinary disorders) | 11 (20)
Pulmonary event (Respiratory, thoracic and mediastinal disorders) | 5 (14)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 12 (35)
Leukocytes (Blood and lymphatic system disorders) | 19 (66)
Lymphopenia (Blood and lymphatic system disorders) | 17 (63) — Grade 1-3
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 5 (7)
Platelets (Blood and lymphatic system disorders) | 14 (28)
Palpitation (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 7 (14)
Fatigue (General disorders) | 18 (57)
Weight change (General disorders) | 4 (9)
Coagulation (Investigations) | 1 (2)
Dermatologic symptoms (Skin and subcutaneous tissue disorders) | 14 (28)
Nausea (Gastrointestinal disorders) | 10 (18)
Other Gastrointestinal event (Gastrointestinal disorders) | 14 (60)
Hemorrhage (General disorders) | 9 (31)
Infection (Infections and infestations) | 6 (8)
Edema (General disorders) | 5 (11)
Gynecologic symptoms (Reproductive system and breast disorders) | 4 (5)
Pain (General disorders) | 15 (42)
Mood Alteration (Psychiatric disorders) | 5 (7)
Neurological event (Nervous system disorders) | 8 (16)
Musculoskeletal event (Musculoskeletal and connective tissue disorders) | 3 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 18 (44)
Other metabolic/laboratory (Metabolism and nutrition disorders) | 19 (125)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes